CLINICAL TRIAL: NCT00010751
Title: Chronic Diabetic Painful Neuropathy and Cardiovascular Risk Factors in NIDDM: An Alternative Approach.
Brief Title: Effects of Reiki on Painful Neuropathy and Cardiovascular Risk Factors
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Allocation: Randomized | Masking: Single | Purpose: Treatment
Other Study IDs: P50 AT000011-1; P50AT000011 (NIH); NCT00009412 (obsolete NCT alias)
Record Dates: First submitted 2001-02-02; First posted 2001-02-05 (Estimated); Last update posted 2006-08-18 (Estimated); Status verified 2006-08

CONDITIONS: Coronary Disease; Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Coronary Disease; Diabetes Mellitus, Type 2 | interventions — Therapeutic Touch

INTERVENTIONS:
Procedure: Reiki

SUMMARY:
The object of this study is to determine if Reiki will improve glycemic control and cardiac autonomic function diabetic patients with painful neuropathy.

DETAILED DESCRIPTION:
The incidence of coronary heart disease(CHD) in type II diabetes is currently at least 20% in subjects 65 years and older. Numerous data suggest that hyperglycemia may be an independent risk factor for macrovascular complications. Diabetic painful neuropathy (DPN) affects 5-50% of patients with diabetes and is exacerbated by poor glycemic control. DPN is characterized by acute functional abnormalities in nerve fibers followed by chronic nerve fiber loss and blunted nerve fiber regeneration. Symptoms include tingling and burning sensations in the calves, ankles and feet. Pharmacological treatment of diabetic autonomic neuropathy (DAN) and DPN include tricyclic antidepressants, which are cardiotoxic and have a low efficacy rate. The ADA recommends the utilization of diet and exercise as the primary means of glycemic control, and therefore of DPN. Because of the increased levels of extremity pain, patients with DPN are less likely to include exercise as a part of their health regimen. Diabetic autonomic neuropathy (DAN) commonly complicates diabetes and has been invoked as a cause of sudden death in diabetic patients. The excess cardiac mortality in diabetics appears to be augmented by the presence of DAN in patients with advanced deficits in sympathetic cardiovascular enervation which may augment cardiac arrhythmogenesis. An bio-energy modality known as Reiki is an energy manipulation technique similar to Therapeutic Touch, a hands-on modality familiar in nursing for the relief of chronic pain, as well as accelerate healing in full thickness dermal wounds. The study approach is to apply Reiki to patients with DPN +/- DAN in a semi-double blind, randomized, crossover study to ascertain if glycemic control and cardiac autonomic function are improved in these patients. Outcome measures will include HBA1c values, the McGill-Melzack Pain Questionnaire, and a quality of life questionnaire. Participants will also be tested as to their ability to tolerate exercise by a 6 minute walk test. This study will help elucidate whether an bio-energy technique can reduce pain levels, improve glycemic control by increasing exercise tolerance and improve cardiac autonomic function, both major contributors to CHD mortality.

ELIGIBILITY:
* NIDDM as defined by the World Health Organization
* Diagnosed with DPN +/- DAN for a duration of no less than six months
* Women of childbearing potential must be using an acceptable method of contraception to prevent pregnancy when they are enrolled in the study and must agree to continue to practice an acceptable method of contraception for the duration of their participation
* Stability of diabetes control by documentation of <1% fluctuation of HbA1c levels over the last twelve months and 3 or less mild hypoglycemic reactions per week. All subjects must be prepared to monitor blood glucose values three to four times daily
* HbA1c should be <10%
* Ability to give informed consent and willingness to sign the Institutional Review Board approved consent form
* Willingness to cooperate with medical therapy and follow up for the 12 months of the study duration
* Have the ability to understand English

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 1998-09; Study Completion 2004-06

CONTACTS AND LOCATIONS:
Overall Officials: Martin Stevens, MD, Principal Investigator — University of Michigan
Locations (1):
- Taubman Center, Ann Arbor, Michigan, United States